CLINICAL TRIAL: NCT07108400
Title: Efficacy of a Combination of Ultrasound-guided Intra-articular Injections of Hyaluronic Acid, High-power Laser Therapy and Rehabilitation on Functioning in Patients Affected by Hip Osteoarthritis: a Randomized Controlled Trial
Brief Title: Efficacy of a Combination of Ultrasound-guided Intra-articular Injections of Hyaluronic Acid, High-power Laser Therapy and Rehabilitation on Functioning in Patients Affected by Hip Osteoarthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: De Sire Alessandro (Other)
Responsible Party: Sponsor-Investigator, De Sire Alessandro, professor, University of Catanzaro
Organization: University of Catanzaro (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 429/2021
Record Dates: First submitted 2025-06-13; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hip Osteoarthritis
Keywords: lasertherapy; hyaluronic acid; hip osteoarthritis; functioning; rehabilitation; pain
MeSH Terms: conditions — Osteoarthritis, Hip; Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental)
  Interventions: Procedure: ultrasound-guided injections of hyaluronic acid plus high-power laser therapy
- Control group (Sham Comparator)
  Interventions: Procedure: ultrasound-guided injections of hyaluronic acid plus sham" high-power laser therapy

INTERVENTIONS:
Procedure: ultrasound-guided injections of hyaluronic acid plus high-power laser therapy — Received two ultrasound-guided injections of hyaluronic acid into the coxo-femoral joint, 10 sessions of physical therapy specifically targeting hip OA (5 sessions/week for two weeks) lasting 45 minutes, and 10 sessions of active high-power laser therapy using a diode laser.
  Arms: Study group
Procedure: ultrasound-guided injections of hyaluronic acid plus sham" high-power laser therapy — Received two ultrasound-guided injections of hyaluronic acid into the coxo-femoral joint, 10 sessions of physical therapy specifically targeting hip OA (5 sessions/week for two weeks) lasting 45 minutes, and 10 sessions of "sham" high-power laser therapy using a diode laser, due to the presence of a light pointer and an acoustic signal of the device, which made it impossible to distinguish the active treatment from the sim-ulated one.
  Arms: Control group

SUMMARY:
High-power laser therapy (HPLT) is effective in treating musculoskeletal conditions, reducing pain and improving joint functionality. This randomized controlled trial (RCT) aimed to explore the effectiveness of a combination of HPLT, hyaluronic acid injections, and rehabilitation for patients with hip osteoarthritis.

DETAILED DESCRIPTION:
This RCT enrolled adults over 18 with a diagnosis of hip osteoarthritis (stages 1-3) who experience hip pain of 4 or higher on a scale. Participants must have a BMI under 30. Patients were randomly assigned to either a study or control group, with both patients and assessors blinded to the treatment. The study group received hyaluronic acid injections, physiotherapy, and active HPLT, while the control group received the same management, except for sham HPLT. We used the Harris Hip Score (HHS) as primary outcome to assess hip function-ing, and as secondary outcomes the following ones: Numeric Rating Scale (NRS) for pain, Eu-roQoL (EQ-5D) for quality of life, and the 6-minute walking test for physical performance. Eval-uations were conducted at multiple timepoints: baseline (T0), post-treatment (T1), and follow-ups at 3 months (T2), 6 months (T3), and 12 months (T4) after the first visit. 57 patients were ran-domly assigned to either a study group (28 patients) or a control group (29 patients).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Diagnosis of hip OA (stage ≤ 3 according to the Kellgren and Lawrence classification)
* Hip pain assessed with the Numeric Rating Scale ≥ 4
* Body mass index (BMI) less than 30 kg/m²
* Suspension of anti-inflammatory drugs (NSAIDs), opioids, corticosteroids, muscle relaxants or any other therapy that could interfere with the study assessments.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score < 24
* Concurrent treatment with an-ti-inflammatory drugs or rehabilitation therapies; Rheumatoid arthritis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
the Harris Hip Score (HHS) | - T0: Baseline ; - T1: 2 week from the baseline ; - T2: 3 months from the baseline; - T3: 6 months from the baseline; - T4: 12 months from the baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University "Magna Graecia "of Catanzaro, Catanzaro, CZ
  - University "Magna Graecia "of Catanzaro, Catanzaro

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT07108400/Prot_SAP_ICF_000.pdf